CLINICAL TRIAL: NCT05053217
Title: Effect of Fibromyalgia on Outcomes of Transforaminal Epidural Steroid Injection Treatment in Lumbar Radicular Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2021.685
Record Dates: First submitted 2021-09-16; First posted 2021-09-22 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-09

CONDITIONS: Herniated Disk Lumbar; Fibromyalgia
Keywords: fibromyalgia; lumbar disc herniation; tfese
MeSH Terms: conditions — Fibromyalgia; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients diagnosed with fibromyalgia (Active Comparator)
  Interventions: Procedure: transforaminal epidural steroid injection
- Patients without a diagnosis of fibromyalgia (Active Comparator)
  Interventions: Procedure: transforaminal epidural steroid injection

INTERVENTIONS:
Procedure: transforaminal epidural steroid injection — In the transforaminal approach, a small amount of drug is injected into the epidural space, and in previous studies, reduction in pain and improvement in functionality were found in patients with lumbar radicular pain in the short and medium term.

SUMMARY:
Lumbar radicular pain is defined as low back and leg pain caused by inflammation in the affected nerve root due to various etiological factors. In its treatment, there are various options such as anti-inflammatory drugs, physical therapy modalities, exercises, epidural steroid injections, and surgery. Epidural steroid injections have also become a frequently applied method in the treatment of lumbar radicular pain unresponsive to conservative treatments. The steroid applied here acts by suppressing the inflammation around the affected nerve root. Epidural steroid injections can be applied in lumbar radicular pain with 3 different approaches: caudal, interlaminar and transforaminal. In the transforaminal approach, a small amount of drug is injected into the epidural space, and in previous studies, reduction in pain and improvement in functionality were found in patients with lumbar radicular pain in the short and medium term. As far as we know, there is no previous study investigating the effect of fibromyalgia on TFESE treatment outcomes. For this reason, the aim of our study is to examine the effect of fibromyalgia on treatment outcomes in patients who underwent TFESE for lumbar radicular pain.

ELIGIBILITY:
Inclusion Criteria:

* Findings of root compression on MRI, lumbar radicular pain for at least 3 months, no previous history of lumbar spinal surgery, pain score of 4 and above according to the numerical rating scale (NRS), and ACR 2016 diagnostic criteria for the fibromyalgia group were met. patients

Exclusion Criteria:

* Patients who received lumbar epidural steroid injection in the last 3 months, who have pregnancy-breastfeeding, bleeding diathesis, contrast hypersensitivity, and patients who did not give consent for participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Successful Response | 3 months
  The primary outcome measure of our study is successful response (>50% reduction in NRS)

SECONDARY OUTCOMES:
Numerical Rating Scale | 3 months
  Numerical rating scale (NRS) is used to convert some values into numeric values that cannot be evaluated numerically
Istanbul Low Back Pain Disability Index (ILBPDI) | 3 months
  Istanbul Low Back Pain Disability Index (ILBPDI) is a scale developed to evaluate functional disability in patients with chronic low back pain, scoring 18 subjects
Short Form 12 (SF-12) | 3 months
  Short Form 12 (SF-12) is a quality of life assessment scale consisting of 8 sub-dimensions and 12 items

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No